CLINICAL TRIAL: NCT01981616
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Single Dose Study in Healthy Subjects to Determine the Immune Response to Systemic and Mucosal Antigenic Challenge in the Presence of Vedolizumab
Brief Title: Immune Response to Systemic and Mucosal Antigenic Challenge in the Presence of Vedolizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C13013; 2011-001874-24 (EudraCT Number); U1111-1147-3216 (Registry Identifier: WHO)
Record Dates: First submitted 2013-10-30; First posted 2013-11-11 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: Drug therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — vedolizumab; LDP-02; Hepatitis B Vaccines; Cholera Vaccines; Dukoral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vedolizumab 750 mg (Experimental): Vedolizumab 750 mg, intravenous (IV) infusion, once on Day 1. Also 3 doses of a hepatitis B vaccine series on Days 4, 32 and 60, and 2 doses of an oral cholera vaccine on Days 4 and 18.
  Interventions: Drug: Vedolizumab; Biological: Hepatitis B vaccine; Biological: Oral cholera vaccine
- Placebo (Placebo Comparator): Vedolizumab placebo-matching, IV infusion, once on Day 1. Also 3 doses of a hepatitis B vaccine series on Days 4, 32 and 60, and 2 doses of an oral cholera vaccine on Days 4 and 18.
  Interventions: Drug: Placebo; Biological: Hepatitis B vaccine; Biological: Oral cholera vaccine

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab for intravenous infusion
  Other Names: Entyvio; MLN0002; MLN02; LDP-02
  Arms: Vedolizumab 750 mg
Drug: Placebo — Placebo intravenous infusion
  Arms: Placebo
Biological: Hepatitis B vaccine
  Other Names: HBVAXPRO
Biological: Oral cholera vaccine
  Other Names: Dukoral

SUMMARY:
The primary purpose of this study is to determine the rates of seroconversion to a hepatitis B vaccine series after a single 750 mg intravenous (IV) dose of vedolizumab or placebo. Secondary objectives are to determine the rates of seroconversion to an oral cholera vaccine series, assess change in anti-hepatitis B surface antibodies and assess the safety and tolerability of a single 750-mg IV dose of vedolizumab.

ELIGIBILITY:
Inclusion criteria

1. Male or female participants 18 to 39 years of age.
2. Body mass index (BMI) between 18 and 32 kg/m^2, inclusive.
3. Females who: are postmenopausal for at least 1 year before the Screening visit, OR; are surgically sterile, OR; if they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
4. Males, even if surgically sterilized (ie, status postvasectomy), who: agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or; agree to completely abstain from heterosexual intercourse.
5. Is willing and able to provide written informed consent and to comply with all study requirements.
6. Has suitable venous access for the study-required infusions and blood samples.

Exclusion criteria

1. Known exposure to hepatitis B virus.
2. Known prior hepatitis B vaccination, irrespective of number of doses received, or any previous employment in a healthcare setting.
3. Seropositivity for prior hepatitis B infection or hepatitis B vaccination during the Screening period.
4. Known exposure to cholera or prior Dukoral exposure, irrespective of number of doses received.
5. History of major cardiovascular, pulmonary, hepatic, renal, gastrointestinal (GI), genitourinary, hematological, immunological, psychiatric, or other major medical disorder.
6. History of any major neurological disorder, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease, or any neurological disorders that would confound neurological examination, or results of the subjective or objective progressive multifocal leukoencephalopathy (PML) checklist during the study.
7. Any history of coagulation disorders, or history or current use of anticoagulation therapy (eg, warfarin, heparin).
8. Any disorder that requires chronic or regular use of any form of corticosteroid (including but not limited to topical, intranasal, rectal, etc), immunomodulator (eg, azathioprine) therapy, or other immunosuppressant (eg, mycophenolate, tacrolimus, tumor necrosis factor-alpha (TNF-α) antagonist).
9. Regular use of herbal, homeopathic or natural supplements including but not limited to putative immune stimulants. Participants must not have used any of these agents within 30 days of enrollment.
10. Female participants who are lactating or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 predose; women considering becoming pregnant while on study are to be excluded.
11. Acute illness within the preceding 30 days that, in the opinion of the investigator, could pose a threat or harm to the participant or obscure laboratory test results or interpretation of data on exposure to vedolizumab (eg, mononucleosis).
12. Any history of malignancy, except for the following: (a) adequately-treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to enrollment; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years before enrollment.
13. Had a surgical procedure requiring general anesthesia within 30 days before the initial Screening visit or is planning to undergo a surgery that requires general anesthesia during the study period. Minor surgeries that are medically necessary and that do not require general anesthesia may be allowable during the study period.
14. One or more positive responses on the PML subjective symptom checklist at screening or before dosing on Day 1.
15. Blood donation within 60 days before screening.
16. Unable to attend all study days or comply with protocol requirements.
17. Any other reason that, in the opinion of the investigator, would confound the conduct of this study or the interpretation of the results.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- ICON Development Solutions, Manchester, United Kingdom

REFERENCES:
- [Derived] Wyant T, Leach T, Sankoh S, Wang Y, Paolino J, Pasetti MF, Feagan BG, Parikh A. Vedolizumab affects antibody responses to immunisation selectively in the gastrointestinal tract: randomised controlled trial results. Gut. 2015 Jan;64(1):77-83. doi: 10.1136/gutjnl-2014-307127. Epub 2014 Apr 24. PMID 24763133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United Kingdom from 13 September 2011 to 13 July 2012.
Pre-assignment Details: Healthy participants were randomized in a 1:1 ratio to receive a single dose of placebo or vedolizumab.
Groups:
- Vedolizumab 750 mg: Vedolizumab 750 mg solution, intravenous (IV) infusion, once on Day 1. Also 3 doses of a hepatitis B vaccine series on Days 4, 32 and 60, and 2 doses of an oral cholera vaccine on Days 4 and 18.
- Placebo: Vedolizumab placebo-matching solution, IV infusion, once on Day 1. Also 3 doses of a hepatitis B vaccine series on Days 4, 32 and 60, and 2 doses of an oral cholera vaccine on Days 4 and 18.
Period: Overall Study
Arm/Group | Vedolizumab 750 mg | Placebo
Started | 64 | 63
Completed | 63 | 62
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vedolizumab 750 mg | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.64) | 27.3 (5.33) | 27.5 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 44 | 43 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  White | 62 | 56 | 118
  Black | 1 | 1 | 2
  Asian | 1 | 2 | 3
  Other | 0 | 4 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 64 | 62 | 126
Region of Enrollment [Number; unit: participants]
  United Kingdom | 64 | 63 | 127
Height [Mean (Standard Deviation); unit: cm] | 173.4 (8.89) | 173.1 (7.94) | 173.3 (8.40)
Weight [Mean (Standard Deviation); unit: kg] | 75.0 (13.48) | 76.2 (11.53) | 75.6 (12.51)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (3.34) | 25.4 (2.71) | 25.1 (3.04)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Immune Response to Hepatitis B Vaccine at Day 74
Description: Immune response was defined as hepatitis B surface antibody (anti-HBs) ≥ 10 IU/L.
Time Frame: Day 74
Population: The Per Protocol Population consisted of all participants who received any amount of study drug and who met predefined evaluability criteria, including receiving the correct and complete dose of study drug, completed both Baseline and day 72 serology assessments and full schedule of hepatitis B vaccine and immunomodulator or corticosteroid use.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 750 mg | Placebo
Number analyzed (Participants) | 61 | 62
percentage of participants | 88.5 [80.5 to 96.5] | 90.3 [83.0 to 97.7]
Statistical Analysis 1: Comparison: Vedolizumab 750 mg vs Placebo; Test type: Non-Inferiority or Equivalence — With 55 evaluable participants in each group, the study would have at least 80% power to exclude the non-inferiority margin of 15% with the lower bound of the 1-sided 95% confidence interval (CI) on the difference in proportions between vedolizumab- and placebo-treated participants, assuming a 90% seroconversion rate (anti-HBs of 10 IU/L) for hepatitis B vaccine. If the lower bound of this interval was less than -15% (ie, more negative), then the null hypothesis was accepted; Difference from placebo = -1.8, 95% CI 2-sided [-12.7 to 9.1]

2. Secondary Outcome: Percentage of Participants With an Immune Response to Oral Cholera Vaccine
Description: A positive immune response was defined as an increase of greater than 4-fold over the Baseline immunoglobulin M (IgM), IgG, or IgA anticholera antibodies.
Time Frame: Baseline and Day 74
Population: The Dukoral Population was defined as all participants who had evaluable samples for assessing immune response to cholera vaccine (Dukoral) vaccine at any visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 750 mg | Placebo
Number analyzed (Participants) | 63 | 62
percentage of participants | 82.5 [73.2 to 91.9] | 96.8 [92.4 to 100.0]
Statistical Analysis 1: Comparison: Vedolizumab 750 mg vs Placebo; Test type: Non-Inferiority or Equivalence — The sample size of 55 evaluable subjects in the vedolizumab 750 mg IV group and 55 evaluable participants in the placebo group provided at least 71% power to exclude the non-inferiority margin of 15% with the lower bound of the 1-sided 95% CI on the difference in proportions between vedolizumab- and placebo-treated participants, assuming an 85% seroconversion rate to the oral cholera vaccine (Dukoral); Difference from placebo = -14.2, 95% CI 2-sided [-24.6 to -3.9]

3. Secondary Outcome: Anti-Hepatitis B Surface Antibody Over Time
Time Frame: Baseline and Days 18, 32, 60 and 74
Population: Per Protocol Population; "n" indicates the number of participants with available data at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/L
Arm/Group | Vedolizumab 750 mg | Placebo
Number analyzed (Participants) | 61 | 62
IU/L
  Baseline (n=24, 31) | 1.2 (51.9) | 1.0 (12.5)
  Day 18 (n=39, 40) | 2.5 (501.0) | 1.3 (73.5)
  Day 32 (n=37, 41) | 2.3 (472.8) | 1.6 (99.9)
  Day 60 (n=58, 59) | 16.3 (501.3) | 15.2 (365.8)
  Day 74 (n=59, 62) | 129.6 (359.3) | 114.4 (539.6)

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a subject administered a pharmaceutical product; the untoward medical occurrence did not necessarily have a causal relationship with this treatment.
  Serious adverse event (SAE) meant any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of an existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly/birth defect or was a medically important event. Relationship of each AE to study drug was determined by the Investigator.
Time Frame: From the first dose of study medication through Day 127
Population: The Safety Population was defined as all participants who received any amount of study drug (vedolizumab or placebo) based on what they actually received.
Measure: Number; unit: participants
Arm/Group | Vedolizumab 750 mg | Placebo
Number analyzed (Participants) | 64 | 63
participants
  Any adverse event | 41 | 50
  Drug-related adverse event | 22 | 22
  Adverse event resulting in study discontinuation | 0 | 1
  Serious adverse event | 0 | 1
  Serious infection adverse events | 0 | 0
  Drug-related serious adverse event | 0 | 0
  Serious adverse event resulting in discontinuation | 0 | 0
  Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through Day 127.
Arm/Group | Vedolizumab 750 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/63
Other Adverse Events (participants affected / at risk) | 24/64 | 25/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 750 mg (N=64) | Placebo (N=63)
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 750 mg (N=64) | Placebo (N=63)
Viral upper respiratory tract infection (Infections and infestations) | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Gastroenteritis (Infections and infestations) | 2 | 5
Headache (Nervous system disorders) | 12 | 8
Nausea (Gastrointestinal disorders) | 4 | 0
Fatigue (General disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other